CLINICAL TRIAL: NCT01242449
Title: A Phase II Investigation of Oral Vinorelbine in Combination With Trastuzumab for 1st and 2nd Line Treatment of Women With Metastatic HER2 Positive Breast Cancer
Brief Title: Oral Vinorelbine in Combination With Trastuzumab for Metastatic Breast Cancer
Acronym: OVINTRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2010-021618-42
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Metastatic; HER2 positive; vinorelbine
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Trastuzumab; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Trastuzumab — Initial dose 8 mg/kg i.v. Subsequently, 6 mg/kg i.v. at intervals of 3 weeks
Drug: Vinorelbine — Initial dose 70 mg/m2 on days 1 and 8 (capsules) If well tolerated, subsequently 90 mg/m2 on days 1 and 8. Capsule on day 1 to be taken at the hospital, and on day 8 at home.

SUMMARY:
This phase II study will investigate oral vinorelbine 90 mg/m2 on days 1 + 8 at 3 weeks intervals in combination with trastuzumab as 1st and 2nd line treatment of women with metastatic HER2 positive breast cancer.

Oral vinorelbine has shown the same overall response rate as i.v. vinorelbine in metastatic breast cancer, and capsules are generally better tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Woman ≥ 18 years of age.
* PS 0-2. Expected lifetime of more than 12 weeks.
* Histologically verified breast cancer(adenocarcinoma)
* Primary tumor or metastasis is HER2 positive with IHC3+ or FISH+ (ratio ≥ 2.2).
* Documented metastatic breast cancer with min. one lesion measureable according to the RECIST 1.1 criteria. All solitary lesions must be verified cytologically/histologically if representing the only evidence of malignancy.
* The patient may have received (neo-) adjuvant chemotherapy (taxanes, anthracyclines and trastuzumab) and 1st line chemotherapy in combination with trastuzumab for metastatic disease.
* The patient may have received previous adjuvant antihormonal treatment for metastatic breast cancer.
* The patient may receive radiation therapy, however, not against lesions used for response evaluation.
* Normal heart function, LVEF ≥ 50% measured by MUGA/EKKO.
* Normal bone marrow function: Hemoglobin ≥ 6 mmol/l, ANC ≥ 1.5x10^9/l. Thrombocytes ≥ 100x10^9/l.
* Normal liver function: Bilirubin ≤ 1.5 x upper normal level, ALAT ≤ 2.5 x upper normal level, BASP ≤ 2.5 x upper normal level (≤ 5 if presence of bone metastases).
* Normal renal function: Creatinine ≤ upper normal level. In case of raised creatinine the measured/calculated GFR must be ≥ 50 ml/min.
* Fertile women must present a negative pregnancy test and use contraceptives during and 3 months after treatment. An IUD without hormone is considered a safe contraceptive.
* Written and orally informed consent prior to any study related procedure.

Exclusion Criteria:

* Local recurrence or counter-lateral breast cancer without other dissemination.
* Pregnant or breastfeeding women.
* Clinical symptoms of CNS metastases, incl. meningeal carcinomatosis.
* Malabsorption syndrome or other disease affecting the gastrointestinal function. Resection of the ventriculus or the small intestine, which can affect absorption of oral vinorelbine.
* Dysphagia or other conditions preventing the patient from swallowing tablets.
* Mental or social conditions preventing treatment or follow-up.
* Serious concurrent medical condition, such as:

  * AMI within 12 months or unstable angina.
  * Heart incompensation NYHA III or IV or uncontrolled hypertension (systolic > 150 mm/hg and/or diastolic >100 mm/hg).
  * Serious arrythmia requiring medication, excl. atrial fibrillation and paroxystic supraventricular tachycardia.
  * Active infection, uncontrolled diabetes or hypercalcemia.
* Other concurrent experimental treatment.
* Concurrent antihormonal treatment of metastatic breast cancer.
* Known neuropathia ≥ grade 2.
* Other previous malignant disease within the past 5 years excl. non-melanoma skin cancer and carcinoma in situ cervicis uteri.
* Previous treatment with vinca alkaloid.
* Previous serious allergic or unexpected reactions to trastuzumab treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | Every 9 weeks. Up to 2 years
  CT scan and MUGA scan

SECONDARY OUTCOMES:
Progression free survival | Every 9 weeks from date of first treatment until progression or death. Up to 2 years
  CT scan
Overall Survival | From date of inclusion until date of death. Up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Troels Bechmann, MD, Principal Investigator — Department of Oncology, Vejle Hospital; Erik H Jakobsen, MD, Study Chair — Department of Oncology, Vejle Hospital
Locations (3):
- Denmark (3):
  - Dept. of Oncology, Aalborg Sygehus, Aalborg
  - Dept. of Oncology, Esbjerg Hospital, Esbjerg
  - Department of Oncology, Vejle Hospital, Vejle